CLINICAL TRIAL: NCT05488665
Title: The COMPLETE Treatment of Bifurcation With Two-stent Techniques: Randomized Comparison of Crush Versus Culotte Technique
Acronym: COMPLETE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2022-0033
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crush technique group (Experimental): Two stenting with the Crush technique
  Interventions: Device: Crush technique
- Culotte technique group (Active Comparator): Two stenting with the Culotte technique
  Interventions: Device: Culotte technique

INTERVENTIONS:
Device: Crush technique — Treatment for bifurcation with the Crush technique
  Arms: Crush technique group
Device: Culotte technique — Treatment for bifurcation with the culotte technique
  Arms: Culotte technique group

SUMMARY:
In this COMPLETE randomized trial, using the contemporary second-generation drug-eluting stent, we aimed to test whether the crush technique is superior to the culotte technique for the treatment of bifurcation lesions in terms of 1-year target-lesion failure.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥19 years
2. De novo coronary lesions eligible for drug-eluting stent implantation
3. Medina 1,1,1 or 1,0,1 or 0,1,1 de novo bifurcation lesions (LM or non-LM) and those of main vessel or side branch can be covered by 2 stents
4. Reference vessel diameter of side branch ≥2.5 mm by visual estimation

Exclusion criteria

1. Current or potential pregnancy
2. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
3. Subjects with ST elevation myocardial infarction <24 h from the onset of chest pain
4. Cardiogenic Shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-09-27 (Estimated); Study Completion 2028-09-27 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  The composite of cardiovascular death, target vessel myocardial infarction or clinically driven target lesion revascularization

SECONDARY OUTCOMES:
Cardiovascular death | 1 year
  Death resulting from cardiovascular causes.
Target vessel myocardial infarction | 1 year
  The definition of myocardial infarction followed the fourth universal definition of myocardial infarction and The Academic Research Consortium-2 Consensus Document.
Clinically driven target-lesion revascularization | 1 year
  a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
All-cause of death | 1 year
Target-vessel or non-target vessel myocardial infarction | 1 year
  The definition of myocardial infarction followed the fourth universal definition of myocardial infarction and The Academic Research Consortium-2 Consensus Document.
Definite or probable stent thrombosis | 1 year
  Stent thrombosis is defined according to the Academic Research Consortium definition

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, MD, PhD, Principal Investigator — Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided